CLINICAL TRIAL: NCT06086769
Title: Impact of High Flow Oxygen Therapy on Diaphragm Thickening Fraction in Healthy Subjects. A Prospective Cohort Study
Brief Title: High Flow Oxygen Therapy Effect on Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Principal investigator, Argentinian Intensive Care Society
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: CRIHB #1220 PRISA No. 6256
Record Dates: First submitted 2023-09-29; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers; Diaphragm; Respiratory Rate
Keywords: High flow nasal canula; High flow nasal canula therapy; Diaphragm thickening fraction; Work of breathing; Respiratory rate
MeSH Terms: interventions — Respiratory Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High flow nasal canula — Measurement of diaphragm thickening fraction, respiratory rate and esophageal pressure swing with calculation of diaphragmatic pressure-time product without the use of HFNC and with the use of HFNC at 20 and 40 Liters per minute
  Other Names: diaphragm thickening fraction; esophageal pressure swing; Respiratory rate

SUMMARY:
The use of high-flow nasal cannula (HFNC) has increased. Diaphragmatic ultrasonography is a tool that, as a noninvasive complement to esophageal pressure (Pes) measurement, allows the evaluation of diaphragm function and reflects, through the diaphragm thickening fraction (DTf), the magnitude of diaphragmatic fiber recruitment. The objective of this study was to evaluate the impact of HFNC therapy on the DTf in healthy subjects. Second, this study aimed to assess the behavior of the respiratory rate (RR) and the work of breathing in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects over 18 years old

Exclusion Criteria:

* contraindication for esophageal balloon placement
* diagnosis of lung disease
* smokers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Diaphragm thickening fraction. | Immediately after 5 min of each condition (baseline, 20 and 40 liters per minute) the diaphragmatic thickness was measured at the end of inspiration y de la expiration during 3 consecutive respiratory cycles (each cycle is between 3 and 10 seconds)
  ultrasound measurements were performed by an expert operator (the same in all cases). The ultrasound measurement was performed using a high-resolution linear transducer in real-time in B-mode.
  The diaphragm thickness was measured at the end of expiration and the end of inspiration of the same ventilatory cycle and the average value of 3 ventilatory cycles was recorded. A 2-minute washout period was allowed between each test condition to avoid the summation of effects.
  The DTf and PTPes/min were calculated for each subject in each available condition (baseline - without flow- , wtih 20 and 40 liters per minute):
  DTf = End Inspiratory Diaphragm thickening - End Expiratory Diaphragm thickening / End Expiratory Diaphragm thickening x 100

SECONDARY OUTCOMES:
Respiratory Rate | The number of breaths per minute was recorded in 60 seconds.
  The number of breaths per minute was recorded in 60 seconds.
Esophageal pressure swing (Pes). | 5 minutes each condition
  Difference between basal Pes and maximum inspiratory Pes deflection.
Esophageal pressure-time product per minute (PTPes/min). | Through study completion, an average of 24 weeks
  It was calculated as the area determined by esophageal deflection multiplied by respiratory rate. An ad hoc software developed in MATLAB R2018b (The MathWorks, Inc. Massachusetts, United States) was used for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A Plotnikow, RT, Study Chair — Hospital Británico de Buenos Aires
Locations (1):
- Hospital Britanico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes